CLINICAL TRIAL: NCT03079752
Title: The Prenatal/Early Infancy Project: An Adolescent Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UColorado
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Behavior, Adaptive
MeSH Terms: conditions — Behavior | interventions — Mass Screening; Transportation; Parturition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors were not given access to the participants' original treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Developmental Screening (Active Comparator): Participants received sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age.
  Interventions: Behavioral: Developmental Screening
- Screening plus Transportation (Active Comparator): Participants received sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age; their mothers received free transportation for regular prenatal and well-child care (through child age two).
  Interventions: Behavioral: Developmental Screening; Behavioral: Screening plus Transportation
- Screening, Transport, Prenatal Visits (Active Comparator): Participants received sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age; their mothers received free transportation for regular prenatal and well-child care (through child age two), plus nurse home visiting during pregnancy.
  Interventions: Behavioral: Developmental Screening; Behavioral: Screening plus Transportation; Behavioral: Screening, Transport, Prenatal Visits
- Screen, Transport, Prenatal/Inf Visits (Experimental): Participants received regular sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age; their mothers received free transportation for regular prenatal and well-child care (through child age two), plus nurse home visiting during pregnancy and through child age two.
  Interventions: Behavioral: Developmental Screening; Behavioral: Screening plus Transportation; Behavioral: Screening, Transport, Prenatal Visits; Behavioral: Screen, Transport, Prenatal/Inf Visits

INTERVENTIONS:
Behavioral: Developmental Screening — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment of suspected problems at 12 and 24 months of age
Behavioral: Screening plus Transportation — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment for suspected problems at 12 and 24 months of age; their mothers were provided with free transportation for prenatal and well-child care through child age 2.
  Arms: Screen, Transport, Prenatal/Inf Visits; Screening plus Transportation; Screening, Transport, Prenatal Visits
Behavioral: Screening, Transport, Prenatal Visits — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment for suspected problems at 12 and 24 months of age; their mothers were provided with free transportation for prenatal and well-child care through child age 2, and were provided an average of 9 home visits by nurses during pregnancy.
  Arms: Screen, Transport, Prenatal/Inf Visits; Screening, Transport, Prenatal Visits
Behavioral: Screen, Transport, Prenatal/Inf Visits — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment for suspected problems at 12 and 24 months of age; their mothers were provided with free transportation for prenatal and well-child care through child age 2, and were provided an average of 9 home visits by nurses during pregnancy and 23 during the child's first two years of life.
  Arms: Screen, Transport, Prenatal/Inf Visits

SUMMARY:
The Nurse-Family Partnership, a program of prenatal and infancy home visiting by nurses, has been examined in a series of 3 randomized trials since 1977. It has received considerable attention in the scientific and public policy communities for its replicated effects on a variety of maternal and child health outcomes across these 3 trials, including prenatal health, childhood injuries, rates of subsequent pregnancies, inter-birth intervals, as well as its long-term effects on maternal life-course, criminal behavior, and 15-year-olds' criminal and antisocial behavior in the first trial of the program conducted in Elmira, New York.

DETAILED DESCRIPTION:
Although this program produced positive effects on maternal and child health from pregnancy through the child's fourth year of life, its long-term effects remain unexamined. The current study was conducted to determine the extent to which the beneficial effects of the program set in motion early in the life cycle altered the life-course trajectories of the mothers and the children's adaptive functioning through the first child's 15th birthday. This study examines the long-term effects of the program on two domains of maternal functioning: 1) maternal life course (subsequent children, use of welfare, employment, substance abuse, and encounters with the criminal justice system); and 2) perpetration of child abuse and neglect; and two domains of the children's behavior: 1) their functioning in schools, and 2) their criminal and antisocial behavior. The investigators hypothesized that the program effects in these domains of maternal and child functioning, as in earlier phases of the study, would be greater for families in which the mothers experienced a larger number of chronic stressors and had fewer resources to manage the challenges of living in poverty and being a parent.

ELIGIBILITY:
Inclusion Criteria: Must be offspring of mothers who enrolled in Elmira randomized clinical trial of the Nurse-Family Partnership (known as the Prenatal Early Infancy Project) -

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 1994-03-18 (Actual); Primary Completion 1996-09-12 (Actual); Study Completion 1998-04-30 (Actual)

PRIMARY OUTCOMES:
Timing of Subsequent Births - Mothers | 15 years following birth of first child
  Interval in days between birth date of first child and first subsequent child (self-reported)
Months Received Aid to Families with Dependent Children (AFDC) - Mothers | 15-year interval following birth of first child
  Number of months mother received AFDC (self-reported)
Number of Months Employed - Mothers | 15-year interval following birth of first child
  Number of months employed (self-reported)
Substance Abuse - Mothers | 15-year period following birth of first child
  Count of behavioral impairments due to use of substances (self-reported)
Arrests - Mothers | 15-year interval following birth of first child
  Count of arrests (self-reported)
Child Maltreatment Reports - Mothers | 15-year interval following birth of first child
  Count of substantiated reports of child abuse and neglect in which mother was perpetrator (review of records)
Running Away from Home - Children | 15-year interval following birth of first child
  Count of times ran away from home - self-report
Person in Need of Supervision (PIN) - Children | 15-year period following their birth
  Self report of ever having been adjudicated as a PIN
Arrests - Children | 15-year period following birth
  Count of Arrests - self-report

CONTACTS AND LOCATIONS:
Overall Officials: David Olds, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: Yes
The investigators are in the process of archiving the primary data published for this trial with the University of Michigan Consortium for Political and Social Research.

REFERENCES:
- [Result] Olds DL, Eckenrode J, Henderson CR Jr, Kitzman H, Powers J, Cole R, Sidora K, Morris P, Pettitt LM, Luckey D. Long-term effects of home visitation on maternal life course and child abuse and neglect. Fifteen-year follow-up of a randomized trial. JAMA. 1997 Aug 27;278(8):637-43. PMID 9272895
- [Result] Olds D, Henderson CR Jr, Cole R, Eckenrode J, Kitzman H, Luckey D, Pettitt L, Sidora K, Morris P, Powers J. Long-term effects of nurse home visitation on children's criminal and antisocial behavior: 15-year follow-up of a randomized controlled trial. JAMA. 1998 Oct 14;280(14):1238-44. doi: 10.1001/jama.280.14.1238. PMID 9786373